CLINICAL TRIAL: NCT04507529
Title: 'HjertensGlad'.Inequality in Cardiac Rehabilitation Attendance: Peer-mentors as a Feasible Solution
Brief Title: Peer-mentor Support for Older Vulnerable Myocardial Infarction Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Copenhagen (Other)
Collaborators: Velux Fonden (Other); Danish Nurses Organisation (Other); Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Maria Kjøller Pedersen, Assistant Professor, University College Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Alias: 200348
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-mentoring (Experimental): Peer-mentoring
  Interventions: Other: Peer-mentoring

INTERVENTIONS:
Other: Peer-mentoring — Patients (mentees) are matched with a peer-mentor. Throughout the intervention period (24 weeks), the mentee and the mentor will have informal telephone contact and meet face-to face approximately 8 times during the intervention period.

SUMMARY:
BACKGROUND: Advanced treatment regimens have reduced cardiovascular mortality resulting in an increasingly older myocardial infarction (MI) population in need of cardiac rehabilitation (CR) , the majority (74%) is above 60 years. The positive effect of CR is well established; CR reduces cardiovascular mortality, lowers hospital admissions, and improves quality of life among patients with ischemic heart disease. These positive effects of CR has also been established among older patients. The inherent problem lies in the low attendance rate, often below 50%. Several studies, including studies from Denmark, have shown that low participation in CR is most prevalent among older, vulnerable female patients. The notion vulnerable covers patients with low socioeconomic position (SEP), patients with non-western background and patients living alone, as these groups have particularly low CR attendance. Effective interventions aiming at increasing CR attendance among these low attending groups are thus warranted and the current study will seek to address this.

AIM: To test feasibility and acceptability of methods used in a peer-mentor intervention among older female and vulnerable post MI patients.

DESIGN AND METHODS: The study is designed as a one arm feasibility study. Patients (n=20) are recruited by a dedicated research nurse before discharge from the cardiology department at Nordsjællands Hospital. Data is collected at three timepoints, baseline, 12 weeks and 24 weeks. The patients (mentees) are matched with peer-mentors. Peer-mentoring (i.e. mentoring by a person with a similar life situation or health problem as one self) is a low-cost intervention that holds the potential to improve CR attendance and improve physical and psychological outcomes among older patients. Peer-mentors are role models who can guide and support patients overcoming barriers of CR attendance. Peer-mentoring is unexplored in a CR setting among older, female and vulnerable MI patients; establishing the novelty of the current study.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years and diagnosed with MI and referred to CR and female or low SEP or single living or non-western background.

Exclusion Criteria:

* Patients unable to provide written consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Recruitment | Baseline
  Number of patients included from eligible patients
Dropout | 24 weeks
  Number of patients not completing the intervention
Satisfaction with intervention | 12 weeks
  Semi-structured qualitative interviews with patients
Number of contacts | 24 weeks
  Number of contacts between patient and peer-mentor
Content of contacts | 24 weeks
  Content of contacts between patient and peer-mentor will be assessed through open ended question on questionnaire i.e. 'What was the content of your meeting? e.g face-to-face meeting with conversation about everyday life'
CR attendance | 12 weeks
  Measured as 'self-reported CR attendance'
CR attendance | 24 weeks
  Measured as 'self-reported CR attendance'
Change in Health-related Quality of Life | Baseline to 24 weeks
  Measured using the 'HeartQoL' 'Health-related Quality of Life Questionnaire'. Min. score: 0, max score: 42. Higher scores indicating a better outcome.
Change in Self-efficacy | Baseline to 24 weeks
  Measured using the questionnaire 'General self-efficacy scale'. Min score: 10, max score: 40. Higher scores indicating a better outcome
Change in symptoms of anxiety and depression | Baseline to 24 weeks
  Measured using the questionnaire 'The hospital anxiety and depression scale' (HADS). Min. score: 0, max score 42. Lower scores indicating a better outcome
Change in dietary quality | Baseline to 24 weeks
  Measured using the questionnaire 'Heartdiet'. Higher scores indicating a better outcome
Change in physical activity | Baseline to 24 weeks
  Measured using the questionnaire 'Heartdiet'. Higher scores indicating a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Pedersen, Ph.d., Principal Investigator — University College Copenhagen
Locations (2):
- Denmark (2):
  - Nordsjællands Hospital - Frederikssund, Frederikssund
  - Nordsjællands Hospital - Hillerød, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen M, Bennich B, Boateng T, Beck AM, Sibilitz K, Andersen I, Overgaard D. Peer-mentor support for older vulnerable myocardial infarction patients referred to cardiac rehabilitation: single-arm feasibility study. Pilot Feasibility Stud. 2022 Aug 9;8(1):172. doi: 10.1186/s40814-022-01141-w. PMID 35945611